CLINICAL TRIAL: NCT06150976
Title: Modifying Memory and Attention Adaptation Training (MAAT) For Young Adult Childhood Cancer Survivors
Brief Title: MAAT For Young Adult Cancer Survivors
Acronym: MAAT-YACCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Indiana University School of Medicine (Other); St. Jude Children's Research Hospital (Other)
Responsible Party: Principal Investigator, Donna Posluszny, Associate Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC 23-043
Record Dates: First submitted 2023-11-10; First posted 2023-11-30 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Cancer
Keywords: Cancer; cancer survivorship; cancer-related cognitive impairment; CRCI; Cognitive-behavioral therapy; Memory Attention and Adaptation Training
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MAAT-YS Group (Experimental): This group will be treated with the MAAT-YS cognitive-behavioral therapy.
  Interventions: Behavioral: MAAT-YS

INTERVENTIONS:
Behavioral: MAAT-YS — MAAT is an evidence-based cognitive-behavioral therapy composed of eight 45-minute telehealth appointments and an accompanying workbook.

SUMMARY:
The goal of this clinical trial is to pilot-test a modified version of telehealth-delivered Memory and Attention Adaption Training (MAAT) that is tailored to young adult childhood cancer survivors (ages 18-39; MAAT-YS) with cancer-related cognitive impairment (CRCI). MAAT-YS consists of 8 weekly visits (45-minutes in duration) and participants use a survivor workbook and complete homework between visits. Participants in this single-group pilot trial (N=9) will complete online self-report measures of cognitive symptoms, quality of life, treatment satisfaction and a brief online neuropsychological test battery at baseline and post-MAAT-YS timepoints.

DETAILED DESCRIPTION:
The goal of this clinical trial is to pilot-test a modified version of telehealth-delivered Memory and Attention Adaption Training (MAAT) that is tailored to young adult childhood cancer survivors (ages 18-39; MAAT-YS) with cancer-related cognitive impairment (CRCI). MAAT-YS consists of 8 weekly visits (45-minutes in duration) and participants use a survivor workbook and complete homework between visits.

This pilot trial will determine MAAT-YS feasibility, treatment satisfaction and size of effect in self-report and objective measures of neurocognitive function.

Eligible participants will be 9 individuals who were diagnosed with non-central-nervous system (CNS) cancer (including leukemia/lymphoma without known CNS involvement) prior to the age of 18, are at least 1-year from completion of cancer treatment, including chemotherapy.

Participants will complete online self-report measures of cognitive symptoms, quality of life, treatment satisfaction and a brief online neuropsychological test battery at baseline and post-MAAT-YS timepoints.

If successful, further research is planned with a larger, multi-site randomized controlled trial of MAAT-YS.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18-39
2. Diagnosed prior to 18 years of age with non-CNS solid tumor or leukemia/lymphoma without known CNS involvement
3. At least 1 year after completion of treatment including chemotherapy, cancer-free
4. English fluent
5. Memory or other cognitive problems attributed to cancer and/or cancer treatment
6. Score of <10 on the FACT-Cog Impact on Quality of Life Scale
7. Willing to use telehealth with internet access
8. Willing to provide informed consent to participation

Exclusion Criteria:

1. Severe non-cancer brain injury such as severe traumatic brain injury, stroke or toxic injury causing memory impairments;
2. Currently meeting Diagnostic and Statistical Manual-5 (DSM-5) criteria for a severe psychiatric disorder, including substance abuse, mood, anxiety, or psychotic disorders, as assessed by the PRIME-MD;
3. Scoring 3 or below on the 6-item cognitive screen designed to detect severe memory disorders;59
4. Severe uncorrected sensory impairment (severe hearing or visual impairment).

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2025-02-12 (Actual); Primary Completion 2025-09-05 (Actual); Study Completion 2025-09-05 (Actual)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Therapy-Cognitive (FACT-Cog) v.3. Perceived Cognitive Impairments Scale (PCI) | Baseline to Post-Treatment (after 8 weekly telehealth MAAT-YS visits)
  The PCI assesses perceived cognitive function of participants within a timeframe of the previous 7 days. It consists of 18 items with a 5-point Likert-type rating of 0 (Never) to 4 (Several times a day) with a scoring range of 0-72. Scoring instructions indicate items are reverse scored, such that higher scores denote better perceived cognitive function, lower scores, poorer cognitive function.
CNS Vital Signs (CNSVS) Online Neuropsychological Test Battery (1) Verbal Memory (VBM) (recognition memory for words) | Baseline to Post-Treatment (after 8 weekly telehealth MAAT-YS visits)
  CNSVS Verbal Memory (VBM) is a computer-based neuropsychological test of word recognition and memory for words). The test is measured in standard score units (Mean of 100; SD 15). Higher scores denote better cognitive function.
CNS Vital Signs (CNSVS) Online Neuropsychological Test Battery (2) Symbol Digit Coding (SDC) (visual motor processing speed) | Baseline to Post-Treatment (after 8 weekly telehealth MAAT-YS visits)
  CNSVS Symbol Digit Coding (SDC) is a computer-based neuropsychological test of visual motor processing speed. The test is measured in standard score units (Mean of 100; SD 15). Higher scores denote better cognitive function.
CNS Vital Signs (CNSVS) Online Neuropsychological Test Battery (3) Stroop Test (ST) (visual motor reaction time, processing speed and visual discrimination) | Baseline to Post-Treatment (after 8 weekly telehealth MAAT-YS visits)
  CNSVS Stroop Test (ST) is a computer-based neuropsychological test of visual motor reaction time, processing speed and visual discrimination. The test is measured in standard score units (Mean of 100; SD 15). Higher scores denote better cognitive function.
CNS Vital Signs (CNSVS) Online Neuropsychological Test Battery (4) 4-Part Continuous Performance Test (FPCPT) (sustained attention and working memory) | Baseline to Post-Treatment (after 8 weekly telehealth MAAT visits)
  CNSVS 4-Part Continuous Performance Test (FPCPT) is a computer-based neuropsychological test of sustained attention and working memory. The test is measured in standard score units (Mean of 100; SD 15). Higher scores denote better cognitive function.

SECONDARY OUTCOMES:
Functional Assessment of Cancer Therapy-Cognitive (FACT-Cog) v.3. Impact on Quality-of-Life Scale (IQOL) | Baseline to Post-Treatment (after 8 weekly telehealth MAAT-YS visits)
  The IQOL assesses perceived quality of life impact of cognitive symptoms participants experience within a timeframe of the previous 7 days. It consists of 4 items with a 5-point Likert-type rating of 0 (Not at all) to 4 (Very Much) with a scoring range of 0-16. Scoring instructions indicate items are reverse scored, such that higher scores denote better quality of life, lower scores, poorer quality of life.
Cognitive-Symptom-Checklist-Work-21 (CSC-W-21) | Baseline to Post-Treatment (after 8 weekly telehealth MAAT-YS visits)
  The CSC-W-21 is a 21-tem self-report measure of perceived impact of cognitive symptoms on work (occupational)-related tasks. Respondents are asked to indicate "yes" (1 point) or "no" (0 points) to each item. Higher scores, ranging from 0-21, denote more work-related cognitive symptoms.
Metamemory in Adulthood-Anxiety Scale (MIA-A) | Baseline to Post-Treatment (after 8 weekly telehealth MAAT-YS visits)
  The MIA-A is a 14-item scale that uses a 5-point Likert-type rating for each item (1= Disagree Strongly; 5 Agree Strongly) with item 13 reverse scored. Items are summed with higher scores (range from 14-70) denoting more anxiety associated with perceived cognitive problems in daily life.
Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety v.1. - Short Form 4a | Baseline to Post-Treatment (after 8 weekly telehealth MAAT-YS visits)
  The PROMIS Anxiety v.1 Short Form 4a scale evaluates self-reported fearfulness, cognitive focus, and concentration, as well as emotional distress related to worry and feeling uneasy over the past 7 days. It consists of 4 items, each rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a scoring range of 4 to 20. Raw scores are converted to T-scores using PROMIS norms (mean = 50; SD = 10).Raw scores are converted to T-scores using PROMIS norms (mean = 50; SD = 10). Higher scores denote more anxiety.
Patient-Reported Outcomes Measurement Information System (PROMIS) Depression v.1. - Short Form 4a | Baseline to Post-Treatment (after 8 weekly telehealth MAAT-YS visits)
  The PROMIS Depression v.1 Short Form 4a scale evaluates self-reported negative mood, helpless and worthlessness over the past 7 days. It consists of 4 items, each rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a scoring range of 4 to 20. Raw scores are converted to T-scores using PROMIS norms (mean = 50; SD = 10). Higher scores denote more depression.
Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue v.1. - Short Form 4a | Baseline to Post-Treatment (after 8 weekly telehealth MAAT-YS visits)
  The PROMIS Fatigue v.1 Short Form 4a scale evaluates self-reported symptoms of exhaustion, fatigue and interference with daily activity over the past 7 days. It consists of 4 items, each rated on a 5-point scale (1=not at all; 2=a little bit; 3=somewhat; 4=quite a bit; and 5=very much) with a scoring range of 4 to 20. Raw scores are converted to T-scores using PROMIS norms (mean = 50; SD = 10). Raw scores are converted to T-scores using PROMIS norms (mean = 50; SD = 10). Higher scores denote more anxiety.
Patient-Reported Outcomes Measurement Information System (PROMIS) Scale v1.2. Global Health - Physical 2a | Baseline to Post-Treatment (after 8 weekly telehealth MAAT-YS visits)
  The PROMIS Global Health Physical scale is a self-report measure assessing physical health and ability. It consists of 2 items with a 5-point Likert-type rating of 1 (Poor) to 5 (Excellent) with a scoring range of 2-10. Raw scores are converted to T-scores using PROMIS norms (mean = 50; SD = 10). Higher scores denote better physical health.
Patient-Reported Outcomes Measurement Information System (PROMIS) Scale v1.2. Global Health - Mental 2a | Baseline to Post-Treatment (after 8 weekly telehealth MAAT-YS visits)
  The PROMIS Global Health Mental scale is a self-report measure assessing mental health and ability. It consists of 2 items with a 5-point Likert-type rating of 1 (Poor) to 5 (Excellent) with a scoring range of 2-10. Raw scores are converted to T-scores using PROMIS norms (mean = 50; SD = 10). Higher scores denote better mental health.
Credibility/Expectancy Questionnaire (CEQ) | Only administered after Visit 6 of MAAT-YS (after 6 weeks)
  The CEQ is a self-report measure assessing the credibility and expectancy of treatment received. It consists of 6 items, 4 items with a 9-point Likert-type rating of 1 (not at all) to 5 (very much) with a scoring range of 3-27. The other 2 items are on a percentage scale from 0%-100% in increments of 10 with a scoring range of means 0-100%. Higher scores denote higher treatment credibility and expectancy.
Treatment Satisfaction Questionnaire (TSS) | Post-MAAT-YS treatment only (8 weeks)
  The Treatment Satisfaction (TSS) questionnaire is a self-report measure assessing satisfaction of treatment. It consists of 5 items with a 5-point Likert-type rating of 0 (not at all) to 8 (completely) with a scoring range of 0-40 and 1 additional yes/no item about whether traveling for treatment is possible for participation. Higher scores denote more satisfaction with treatment.

OTHER OUTCOMES:
MAAT-YS Fidelity Checklists | Immediately after the 6th visit of the MAAT intervention (6 weeks)
  The MAAT-YS Fidelity Checklists assess the degree to which the MAAT-YS study clinician adheres to specific therapeutic behaviors of the MAAT-YS Clinician Manual. The checklists are administered to 2 independent treatment adherence raters who review randomly selected audio recordings of each of the 8 telehealth-delivered MAAT-YS visits. Behaviors in checklists per each visit are independently rated 0 (no or poor fidelity) to 10 (highest fidelity possible). Rating means are computed for each visit for a score of 0-10 with higher scores denoting higher treatment fidelity.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Ferguson, PhD, Principal Investigator — St. Jude Children's Research Hospital; Donna Posluszny, PhD, Principal Investigator — University of Pittsburgh
Locations (3):
- United States (3):
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Pittsburgh School of Medicine/UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No
There is no data sharing plan with other institutions for this pilot trial.